CLINICAL TRIAL: NCT03984370
Title: Dasiglucagon in the Treatment of Postprandial Hypoglycaemia After Roux-en-Y Gastric Bypass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, MD, professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CKN-DASI-RYGB; 2019-001915-22 (EudraCT Number)
Record Dates: First submitted 2019-06-06; First posted 2019-06-13 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Hyperinsulinemic Hypoglycemia; Postprandial Hypoglycemia
MeSH Terms: conditions — Congenital Hyperinsulinism; Hypoglycemia | interventions — dasiglucagon; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomised, 3-period, 3-treatment, crossover study comprising 3 separate treatment days
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 80 ug of sc dasiglucagon (Experimental): 80 ug of dasiglucagon in a 0.4 mL fluid (saline) is injected abdominal subcutaneous postprandial prior to hypoglycemia.
  Interventions: Drug: ZP4207
- 200 ug of sc dasiglucagon (Experimental): 200 ug of dasiglucagon in a 0.4 mL fluid (saline) is injected abdominal subcutaneous postprandial prior to hypoglycemia.
  Interventions: Drug: ZP4207
- 0.4 mL of sc saline (placebo) (Placebo Comparator): 0.4 mL fluid (saline/placebo) is injected abdominal subcutaneous postprandial prior to hypoglycemia.
  Interventions: Other: Placebo (saline)

INTERVENTIONS:
Drug: ZP4207 — Abdominal SC administration
  Other Names: Dasiglucagon
  Arms: 200 ug of sc dasiglucagon; 80 ug of sc dasiglucagon
Other: Placebo (saline) — Abdominal SC administration
  Arms: 0.4 mL of sc saline (placebo)

SUMMARY:
The aim of this study is investigating the effect of a novel glucagon analogue administration in gastric bypass operated individuals, who are reactive hypoglycemic.

DETAILED DESCRIPTION:
The Roux-En-Y gastric bypass (RYGB) has major health-promoting effects - reversing type-2-diabetes, improving dyslipidemia and inducing robust weight loss. However, several RYGB-individuals, post surgery, suffers from dumping syndrome and postprandial hyperinsulinemic hypoglycemia (PHH) due to the anatomical rearrangement of the gastro-intestinal system. Dasiglugaon (also known as (ZP4207) has shown great pharmacokinetic- and dynamic effects, compared to other glucagon analogues on the market, when administrated to hypoglycemic type-1-diabetics.

Therefore we aim to examine the effects of two different doses of dasiglucagon on the postprandial nadir plasma glucose concentration in RYGB-operated individuals suffering from PHH by use of a mixed meal test (MMT).

The study is designed as a double-blinded, randomised, 3-period, 3-treatment, crossover study comprising 3 separate treatment days in which participants will undergo an MMT along with one of the following double-blinded interventions:

1. Subcutaneous (sc) placebo (saline) injection
2. Sc injection with 80 μg dasiglucagon
3. Sc injection with 200 μg dasiglucagon

ELIGIBILITY:
Inclusion Criteria:

* Documented postprandial hypoglycaemia (<3.9 mmol/l) by 6-day CGM or during a MMT
* Documented plasma glucose concentration excursions >5.0 mmol/l by 6-day CGM or a MMT
* Haemoglobin levels for women >7.3 mmol/l and for men >8.3 mmol/l
* Ferritin >10 μg/l
* Cobalamin >150 pmol/l
* Fasting plasma glucose concentration within the range of 4.0-6.0 mmol/l CKN-DASI-RYGB protocol version 1.0 6
* Normal electrocardiogram (ECG)
* Negative urine human chorionic gonadotropin (hCG) (for fertile women)

Exclusion Criteria:

* Treatment with medication(s) affecting insulin secretion or any antidiabetic drugs
* Treatment with antipsychotics
* Current participation in another clinical trial with administration of investigational drug.
* Previous exposure to dasiglucagon (otherwise known as ZP4207)
* History of liver disease that is expected to interfere with the anti-hypoglycaemic action of glucagon (e.g. liver failure or cirrhosis).
* Pregnancy
* Breastfeeding
* Any factors that, in the opinion of the site principal investigator or clinical protocol chair, would interfere with the safe completion of the study, including medical conditions that may require hospitalization during the trial or allergy to the ingredients in the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Nadir plasma glucose concentration within two hundred forty minutes after MMT | Two hundred forty minutes
  Nadir plasma glucose concentration within two hundred forty minutes after MMT

SECONDARY OUTCOMES:
Time from dasiglucagon administration to recovery (first plasma glucose value above the fasting plasma glucose level | Two hundred forty minutes
  Time from dasiglucagon administration to recovery (first plasma glucose value above the fasting plasma glucose level
Time in hypoglycaemia (plasma glucose concentration <3.9 mmol/l) from study drug administration until 240 minutes | Two hundred forty minutes
  Time in hypoglycaemia
Time below fasting plasma glucose level from study drug administration until two hundred forty minutes | Two hundred forty minutes
  Time below fasting plasma glucose level
Area 1: the area above the glucose curve and below the fasting level from the time of study drug administration until glucose values reach the fasting level. | Two hundred forty minutes
  Area 1
Area 2: the area below the glucose curve and above the fasting level from the time glucose values reach the fasting level until 240 minutes. | Two hundred forty minutes
  Area 2
Edinburgh Hypoglycaemia Symptom Scale (EHSS) responses of the Edinburgh Hypoglycaemia Symptom Scale (EHSS) and early dumping symptoms based on | t=zero to t=Two hundred forty minutes
  likert scale one (absent) to seven (severe)
The Dumping Severity Score (DSS). | t=zero to t=Two hundred forty minutes
  likert scale, zero (absent) to three (severe)
Frequency and severity of adverse events and serious adverse events recorded during the meal test | from t= minus thirty to t=Two hundred forty minutes
  Frequency

CONTACTS AND LOCATIONS:
Overall Officials: Filip M. Knop, Prof., MD, Principal Investigator — Herlev-Gentofte Hospital, Center for Clinical Metabolic Research
Locations (1):
- Center for Clinical Metabolic Research, Herlev-Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen CK, Ohrstrom CC, Kielgast UL, Hansen DL, Hartmann B, Holst JJ, Lund A, Vilsboll T, Knop FK. Dasiglucagon Effectively Mitigates Postbariatric Postprandial Hypoglycemia: A Randomized, Double-Blind, Placebo-Controlled, Crossover Trial. Diabetes Care. 2022 Jun 2;45(6):1476-1481. doi: 10.2337/dc21-2252. PMID 35320361